CLINICAL TRIAL: NCT00717236
Title: A Phase IIIb Multicenter Study With a 12-week Double-blind, Placebo-controlled, Randomized Period Followed by an Open-label, Extension Phase Evaluating Safety/Efficacy of Certolizumab Pegol Given to Patients With Active Rheumatoid Arthritis.
Brief Title: Certolizumab Pegol for the Treatment of Patients With Active Rheumatoid Arthritis
Acronym: REALISTIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C87094; 2008-005427-28 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2012-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Certolizumab pegol; Cimzia; Rheumatoid Arthritis; Joint Disease; Chronic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Joint Diseases | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Certolizumab pegol (CZP) (Experimental)
  Interventions: Drug: Certolizumab pegol (CZP)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Certolizumab pegol (CZP) — 400 mg CZP given as two 200 mg subcutaneous (sc) injections at Weeks 0, 2, and 4, followed by 200 mg CZP given as 1 sc injection on Weeks 6, 8, and 10. At Week 12 subjects enter the open label phase and receive 200 mg of CZP every other week for a minimum 16 additional weeks until CZP is commercially available.
  Other Names: Cimzia
  Arms: Certolizumab pegol (CZP)
Other: Placebo — Placebo (0.9% saline) given as 2 subcutaneous (sc) injections at Weeks 0, 2, and 4, followed by placebo given as 1 sc injection on Weeks 6, 8, and 10. At Week 12 subjects enter the open label phase and receive 200 mg of CZP every other week for a minimum 16 additional weeks until CZP is commercially available.
  Arms: Placebo

SUMMARY:
This is a Phase IIIb multicenter study to evaluate the safety and efficacy of certolizumab pegol (CZP) administered to patients with moderate-to-severe rheumatoid arthritis.

DETAILED DESCRIPTION:
The treatment period starts with a 12-week, double-blind, placebo-controlled, randomized period followed by an open-label extension phase. In the double-blind phase, eligible patients are randomized (4:1 ratio) to receive either certolizumab pegol (CZP) or Placebo up to and including Week 10. The randomization will be stratified according to the three factors: concomitant use of methotrexate (MTX, Yes or No), prior anti-tumor necrosis factor (anti-TNF) use (Yes or No), and disease duration categories (< 2 years or ≥ 2 years). From Week 12 all patients remaining in the study receive open-label CZP for a minimum 16 additional weeks until CZP is commercially available.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with established moderate to severe rheumatoid arthritis

Exclusion Criteria:

* All concomitant diseases or pathological conditions that could interfere and impact the assessment of the study treatment
* Previous clinical trials and previous biological therapy that could interfere with the results in the present clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1648 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (181):
- United States (101):
  - Birmingham, Alabama
  - Montgomery, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Fullerton, California
  - La Jolla, California
  - Los Angeles, California
  - Palm Desert, California
  - Sacramento, California
  - Santa Barbara, California
  - Santa Maria, California
  - Tustin, California
  - Westlake Village, California
  - Whittier, California
  - Denver, Colorado
  - Danbury, Connecticut
  - Trumbull, Connecticut
  - Lewes, Delaware
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Delray Beach, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Orlando, Florida
  - South Miami, Florida
  - Tampa, Florida
  - Tavares, Florida
  - Atlanta, Georgia
  - Coeur d'Alene, Idaho
  - Idaho Falls, Idaho
  - Maywood, Illinois
  - Peoria, Illinois
  - Rock Island, Illinois
  - Springfield, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Louisville, Kentucky
  - Covington, Louisiana
  - Lake Charles, Louisiana
  - Baltimore, Maryland
  - Columbia, Maryland
  - Frederick, Maryland
  - Wheaton, Maryland
  - Boston, Massachusetts
  - Fall River, Massachusetts
  - Battle Creek, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Petoskey, Michigan
  - Duluth, Minnesota
  - Rochester, Minnesota
  - St Louis, Missouri
  - New Brunswick, New Jersey
  - Voorhees Township, New Jersey
  - Albany, New York
  - New York, New York
  - Orchard Park, New York
  - Rochester, New York
  - Roslyn, New York
  - Smithtown, New York
  - Syracuse, New York
  - The Bronx, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Monroe, North Carolina
  - Wilmington, North Carolina
  - Columbus, Ohio
  - Dayton, Ohio
  - Fairfield, Ohio
  - Mayfield, Ohio
  - Oklahoma City, Oklahoma
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - West Reading, Pennsylvania
  - Wexford, Pennsylvania
  - Charleston, South Carolina
  - Jackson, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Lubbock, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Salt Lake City, Utah
  - Newport News, Virginia
  - Richmond, Virginia
  - Spokane, Washington
  - Tacoma, Washington
  - Yakima, Washington
  - Clarksburg, West Virginia
  - Glendale, Wisconsin
  - Milwaukee, Wisconsin
  - Monroe, Wisconsin
- Canada (17):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Rimouski, Quebec
  - Trois-Rivires, Quebec
  - Calgary
  - Mississauga
  - Newmarket
  - Sainte-Foy
- France (13):
  - Amiens
  - Cahors
  - Corbeil-Essonnes
  - Dreux
  - Liévin
  - Montpellier
  - Mulhouse
  - Nantes
  - Orléans
  - Paris
  - Pierre-Bénite
  - Rennes
  - Saint-Priest-en-Jarez
- Germany (25):
  - Bad Neuenahr
  - Baden
  - Berlin
  - Chemnitz
  - Cologne
  - Dresden
  - Duisburg
  - Erfurt
  - Erlangen
  - Freiburg im Breisgau
  - Friedrichroda
  - Goslar
  - Hamburg
  - Hildesheim
  - Hoyerswerda
  - Jena
  - Kiel
  - Leipzig
  - Mainz
  - München
  - Neuss
  - Osnabrück
  - Rostock
  - Wiesbaden
  - Zerbst
- Italy (9):
  - Bologna
  - Genova
  - Iesi
  - Modena
  - Palermo
  - Pisa
  - Prato
  - Siena
  - Udine
- Netherlands (4):
  - Apeldoorn
  - Arnhem
  - Leiden
  - The Hague
- Spain (12):
  - A Coruña
  - Barcelona
  - Madrid
  - Murcia
  - Oviedo
  - Pontevedra
  - Sabadell
  - Salamanca
  - San Cristóbal de La Laguna
  - Santander
  - Santiago de Compostela
  - Torrelavega

REFERENCES:
- [Derived] Smolen JS, Mikuls TR, Galloway J, Muller-Ladner U, Curtis JR, Hashimoto M, Takeuchi T, Choy E, Tanaka Y, Cara C, Lauwerys B, Tilt N, Ufuktepe B, Taylor PC. Do high rheumatoid factor levels impact response to certolizumab pegol in patients with inadequately controlled rheumatoid arthritis? A post hoc analysis of the phase IIIb REALISTIC trial. RMD Open. 2026 Jan 30;12(1):e006094. doi: 10.1136/rmdopen-2025-006094. PMID 41617358
- [Derived] Pope J, Bingham CO 3rd, Fleischmann RM, Dougados M, Massarotti EM, Wollenhaupt J, Duncan B, Coteur G, Weinblatt ME. Impact of certolizumab pegol on patient-reported outcomes in rheumatoid arthritis and correlation with clinical measures of disease activity. Arthritis Res Ther. 2015 Nov 27;17:343. doi: 10.1186/s13075-015-0849-1. PMID 26614481
- [Derived] Weinblatt ME, Fleischmann R, van Vollenhoven RF, Emery P, Huizinga TW, Cutolo M, van der Heijde D, Duncan B, Davies O, Luijtens K, Dougados M. Twenty-eight-week results from the REALISTIC phase IIIb randomized trial: efficacy, safety and predictability of response to certolizumab pegol in a diverse rheumatoid arthritis population. Arthritis Res Ther. 2015 Nov 15;17:325. doi: 10.1186/s13075-015-0841-9. PMID 26568428
- [Derived] Weinblatt ME, Fleischmann R, Huizinga TW, Emery P, Pope J, Massarotti EM, van Vollenhoven RF, Wollenhaupt J, Bingham CO 3rd, Duncan B, Goel N, Davies OR, Dougados M. Efficacy and safety of certolizumab pegol in a broad population of patients with active rheumatoid arthritis: results from the REALISTIC phase IIIb study. Rheumatology (Oxford). 2012 Dec;51(12):2204-14. doi: 10.1093/rheumatology/kes150. Epub 2012 Aug 25. PMID 22923753
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started in July 2008 with subjects from the United States, Canada, France, Germany, Italy, the Netherlands, and Spain. The primary completion date occurred in March 2010, with study completion in March 2011.
Pre-assignment Details: Of the 1648 subjects that were screened, 585 subjects had screen failures. Therefore, 1063 subjects were randomized in this study.
Period: Double-Blind Period
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Started | 851 | 212
Completed | 771 | 184
Not Completed | 80 | 28
Not completed — Adverse Event | 33 | 6
Not completed — Lack of Efficacy | 6 | 6
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 10 | 2
Not completed — Loss of efficacy | 3 | 0
Not completed — Other: Death | 1 | 0
Not completed — Other: Pregnancy | 1 | 0
Not completed — Other: Protocol Violation | 2 | 0
Not completed — Other: Inclusion/Exclusion criteria | 6 | 2
Not completed — Other: Site withdrew | 2 | 0
Not completed — Other: Screening failure | 1 | 0
Not completed — Other: subject withdrew consent | 1 | 1
Not completed — Other: Abnormal chest X-ray | 2 | 1
Not completed — Other: History of adenoid grown | 1 | 0
Not completed — Other: History of cancer | 1 | 0
Not completed — Other: Sponsor request | 1 | 0
Not completed — Other: Inappropriate randomization | 1 | 0
Not completed — Other: Detection of Hepatitis C Virus | 1 | 0
Not completed — Other: Subject moved | 1 | 1
Not completed — Other: Stopped taking DMARD | 1 | 0
Not completed — Other: Prohibited medication taken | 2 | 2
Not completed — Other: Transportation problems | 0 | 1
Not completed — Other: Investigator Decision | 0 | 1
Period: Open-Label Period
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Started | 771 | 184
Completed | 646 | 163
Not Completed | 125 | 21
Not completed — Adverse Event | 29 | 4
Not completed — Lack of Efficacy | 30 | 8
Not completed — Lost to Follow-up | 28 | 4
Not completed — Withdrawal by Subject | 20 | 2
Not completed — Loss of Efficacy | 6 | 1
Not completed — Other: Peripheral Neuropathy | 0 | 1
Not completed — Other: Lack of Compliance | 1 | 1
Not completed — Other: History of Basal Cell Carcinoma | 1 | 0
Not completed — Other: Moved | 1 | 0
Not completed — Other: Investigator Decision | 1 | 0
Not completed — Other: Loss of Staff (unblinded) | 1 | 0
Not completed — Other: Sponsor Request | 3 | 0
Not completed — Other: Cataract Surgery | 1 | 0
Not completed — Other: Administration of Golimumab | 1 | 0
Not completed — Other: Completion Accidently Performed | 1 | 0
Not completed — Other: Medical Monitor Recommendation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Certolizumab Pegol (CZP) | Placebo | Total
Number analyzed (Participants) | 851 | 212 | 1063
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 644 | 164 | 808
  >=65 years | 207 | 48 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (12.43) | 53.9 (12.66) | 55.1 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 660 | 169 | 829
  Male | 191 | 43 | 234
Region of Enrollment [Number; unit: participants]
  France | 14 | 0 | 14
  United States | 575 | 141 | 716
  Canada | 65 | 17 | 82
  Spain | 26 | 8 | 34
  Netherlands | 4 | 0 | 4
  Germany | 154 | 44 | 198
  Italy | 13 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology 20% (ACR20) Response at Week 12
Description: ACR20 responders are subjects with at least 20% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS)
Time Frame: Baseline, Week 12
Population: All 1063 subjects (851 CZP, 212 Placebo) included in the Full Analysis Set (FAS) are included in this analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 851 | 212
percentage of subjects | 51.1 | 25.9

2. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response at Week 12 for Subjects With Concomitant Methotrexate (MTX) Use.
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS), 732 were in the concomitant methotrexate use stratum (589 CZP, 143 Placebo) and are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 589 | 143
percentage of subjects | 52.5 | 28.0

3. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response at Week 12 for Subjects Without Concomitant Methotrexate (MTX) Use.
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS), 331 were in the no concomitant methotrexate use stratum (262 CZP, 69 Placebo) and are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 262 | 69
percentage of subjects | 48.1 | 21.7

4. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response at Week 12 for Subjects With Prior Anti-tumor Necrosis (Anti-TNF) Use
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS), 400 were in the prior anti-tumor necrosis (anti-TNF) use stratum (320 CZP, 80 Placebo) and are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 320 | 80
percentage of subjects | 47.2 | 27.5

5. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response at Week 12 for Subjects Without Prior Anti-tumor Necrosis (Anti-TNF) Use
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS), 663 were in the no prior anti-tumor necrosis (anti-TNF) use stratum (531 CZP, 132 Placebo) and are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 531 | 132
percentage of subjects | 53.5 | 25.0

6. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response at Week 12 for Subjects With Disease Duration < 2 Years
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS), 256 were in the disease duration less than 2 years stratum (206 CZP, 50 Placebo) and are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 206 | 50
percentage of subjects | 50.0 | 30.0

7. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response at Week 12 for Subjects With Disease Duration ≥ 2 Years.
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS), 807 were in the disease duration greater than or equal to 2 years stratum (645 CZP, 162 Placebo) and are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 645 | 162
percentage of subjects | 51.5 | 24.7

8. Secondary Outcome: American College of Rheumatology 50% (ACR50) Response at Week 12
Description: ACR50 responders are subjects with at least 50% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS)
Time Frame: Baseline, Week 12
Population: All 1063 subjects in the Full Analysis Set (FAS) are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 851 | 212
percentage of subjects | 26.6 | 9.9

9. Secondary Outcome: American College of Rheumatology 70% (ACR70) Response at Week 12.
Description: ACR70 responders are subjects with at least 70% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS)
Time Frame: Baseline, Week 12
Population: All 1063 subjects in the Full Analysis Set (FAS) are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 851 | 212
percentage of subjects | 12.9 | 2.8

10. Secondary Outcome: Change From Baseline in DAS28(CRP) [Disease Activity Score-28 (C-reactive Protein)] at Week 12
Description: DAS28(CRP) is calculated using tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/L), and Patient's Global Assessment of Arthritis-Visual Analog Scale (PtGADA-VAS in mm). A lower score indicates less disease activity. Change from baseline is computed as Week 12 value minus baseline value. A negative value in change from baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS) 1037(834 CZP, 203 Placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 834 | 203
units on a scale | -1.70 (1.269) [-6.0 to 1.6] | -0.84 (1.209) [-4.5 to 2.9]

11. Secondary Outcome: Change From Baseline in SDAI (Simplified Disease Activity Index) at Week 12
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/dL), Patient's Global Assessment of Arthritis-Visual Analog Scale (PtGADA-VAS in cm), and Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS in cm). A lower score indicates less disease activity. Change from baseline is computed as Week 12 value minus baseline value. A negative value in change from baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS) 1024 (824 CZP, 200 Placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 824 | 200
units on a scale | -19.66 (14.493) [-69.4 to 30.2] | -10.78 (15.172) [-47.1 to 52.0]

12. Secondary Outcome: Change From Baseline in CDAI (Clinical Disease Activity Index) at Week 12
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Arthritis-Visual Analog Scale (PtGADA-VAS in cm), and Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS in cm). A lower score indicates less disease activity. Change from baseline is computed as Week 12 value minus baseline value. A negative value in change from baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS) 1024 (824 CZP, 200 Placebo) are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 824 | 200
units on a scale | -18.96 (14.019) [-65.8 to 21.2] | -10.93 (14.494) [-47.2 to 43.3]

13. Secondary Outcome: DAS28(CRP) [Disease Activity Score-28 (C-reactive Protein)] Remission (<2.6) at Week 12
Description: DAS28(CRP) is calculated using tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/L), and Patient's Global Assessment of Arthritis-Visual Analog Scale (PtGADA-VAS in mm). A lower score indicates less disease activity.
Time Frame: Week 12
Population: All 1063 subjects in the Full Analysis Set (FAS) are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 851 | 212
percentage of subjects | 16.0 | 5.7

14. Secondary Outcome: SDAI (Simplified Disease Activity Index) Remission (≤3.3) at Week 12
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/dL), Patient's Global Assessment of Arthritis-Visual Analog Scale (PtGADA-VAS in cm), and Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS in cm). A lower score indicates less disease activity.
Time Frame: Week 12
Population: All 1063 subjects in the Full Analysis Set (FAS) are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 851 | 212
percentage of subjects | 7.8 | 1.9

15. Secondary Outcome: CDAI (Clinical Disease Activity Index) Remission (≤2.8) at Week 12
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Arthritis-Visual Analog Scale (PtGADA-VAS in cm), and Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS in cm). A lower score indicates less disease activity.
Time Frame: Week 12
Population: All 1063 subjects in the Full Analysis Set (FAS) are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 851 | 212
percentage of subjects | 8.3 | 1.9

16. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) at Week 12
Description: TJC is calculated based on tenderness response of 28 joints. TJC possible values range from 0 to 28. A lower TJC indicates less joint tenderness. Change from baseline is computed as Week 12 value minus baseline value. A negative value in change from baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS) 1043 (838 CZP, 205 Placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 838 | 205
units on a scale | -7.4 (7.13) [-28 to 18] | -4.5 (7.38) [-28 to 12]

17. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) at Week 12
Description: SJC is calculated based on swelling response of 28 joints. SJC possible values range from 0 to 28. A lower SJC indicates less joint swelling. Change from baseline is computed as Week 12 value minus baseline value. A negative value in change from baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 838 | 205
units on a scale | -6.4 (5.57) [-24 to 13] | -3.6 (5.64) [-21 to 21]

18. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 12
Description: HAQ-DI is derived based on the mean of individual scores in 8 categories of daily living actives (using 20 questions). Each question is scored 0-3 (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do). Change from baseline is computed as Week 12 value minus baseline value. A negative value in change from baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS) 1029 (826 CZP, 203 Placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 826 | 203
units on a scale | -0.38 (0.524) [-2.4 to 1.8] | -0.19 (0.507) [-1.9 to 1.1]

19. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) at Week 12
Description: Change from baseline in CRP (mg/L) is computed as the ratio of Week 12 value divided by baseline value. A ratio less then 1 indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS) 1046 (841 CZP, 205 Placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 841 | 205
mg/L | 0.55 (111.417) [0.0 to 16.6] | 1.05 (89.633) [0.1 to 17.6]

20. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS) at Week 12
Description: Change from Baseline in PAAP-VAS (0 to 100 mm visual analog scale, 0 being no pain and 100 being most severe pain) is computed as Week 12 value minus baseline value. A negative value in change from baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS) 1038 (835 CZP, 203 Placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 835 | 203
mm | -22.1 (28.31) | -10.7 (27.32)

21. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS) at Week 12
Description: Change from Baseline in PtGADA-VAS (0 to 100 mm visual analog scale, 0 being no symptoms and 100 being severe symptoms) is computed as Week 12 value minus baseline value. A negative value in change from baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 835 | 203
mm | -21.5 (27.78) | -10.1 (26.24)

22. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS) at Week 12
Description: Change from Baseline in PhGADA-VAS (0 to 100 mm visual analog scale, 0 being no symptoms and 100 being severe symptoms) is computed as Week 12 value minus baseline value. A negative value in change from baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 12
Population: Of the 1063 subjects in the Full Analysis Set (FAS) 1029 (827 CZP, 202 Placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 827 | 202
mm | -31.2 (23.58) | -19.0 (25.15)

23. Secondary Outcome: Time to Sustained American College of Rheumatology 20% (ACR20) Response
Description: The time from randomization to sustained ACR20 response at 2 consecutive visits (at the latest on Week 12).
Time Frame: Baseline up to Week 12
Population: All 1063 subjects in the Full Analysis Set (FAS) are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 851 | 212
percentage of subjects | 40.4 | 13.2

24. Secondary Outcome: European League Against Rheumatism (EULAR) Response at Week 12
Description: EULAR response (good response, moderate response, or no response) is defined based on the present value and improvement from baseline in DAS28(CRP) [Disease Activity Score-28 (C-reactive protein)].
Time Frame: Baseline, Week 12
Population: All 1063 subjects in the Full Analysis Set (FAS) are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo
Number analyzed (Participants) | 851 | 212
percentage of subjects
  Good response | 28.9 | 10.4
  Moderate response | 44.5 | 37.3
  No response | 26.6 | 52.4

25. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response at Week 28
Description: ACR20 responders are subjects with at least 20% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS). This analysis was carried out using imputation.
Time Frame: Baseline, Week 28
Population: Since imputation was used, all 954 subjects from the Open Label (OL) Set are included in this analysis
Measure: Number; unit: percentage of subjects
Groups:
- Open Label Certolizumab Pegol (CZP): Subjects entering the open label extension at Week 12 receive 200 mg CZP given every other week for a minimum 16 additional weeks until CZP is commercially available.
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 954
percentage of subjects | 58.5

26. Secondary Outcome: American College of Rheumatology 50% (ACR50) Response at Week 28
Description: ACR50 responders are subjects with at least 50% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS). This analysis was carried out using imputation.
Time Frame: Baseline, Week 28
Population: Since imputation was used, all 954 subjects from the Open Label (OL) Set are included in this analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 954
percentage of subjects | 35.0

27. Secondary Outcome: American College of Rheumatology 70% (ACR70) Response at Week 28
Description: ACR70 responders are subjects with at least 70% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS). This analysis was carried out using imputation.
Time Frame: Baseline, Week 28
Population: Since imputation was used, all 954 subjects from the Open Label (OL) Set are included in this analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 954
percentage of subjects | 17.4

28. Secondary Outcome: Change From Baseline in DAS28(CRP) [Disease Activity Score-28 (C-reactive Protein)] at Week 28
Description: DAS28(CRP) is calculated using tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/L), and Patient's Global Assessment of Arthritis-Visual Analog Scale (PtGADA-VAS in mm). A lower score indicates less disease activity. Change from Baseline is computed as the value at Week 28 minus Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was done using a Mixed Effects Repeated Measures Model (MMRM).
Time Frame: Baseline, Week 28
Population: Of the 954 subjects in the Open Label Set (OLS) 840 had observed values at Week 28 and Baseline and are included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 840
units on a scale | -1.94 (0.055)

29. Secondary Outcome: Change From Baseline in SDAI (Simplified Disease Activity Index) at Week 28
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/dL), Patient's Global Assessment of Arthritis-Visual Analog Scale (PtGADA-VAS in cm), and Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS in cm). A lower score indicates less disease activity. Change from Baseline is computed as the value at Week 28 minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was done using a Mixed Effects Repeated Measures Model (MMRM).
Time Frame: Baseline, Week 28
Population: Of the 954 subjects in the Open Label Set (OLS) 828 had observed values at Week 28 and Baseline and are included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 828
units on a scale | -22.35 (0.546)

30. Secondary Outcome: Change From Baseline in CDAI (Clinical Disease Activity Index) at Week 28
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Arthritis-Visual Analog Scale (PtGADA-VAS in cm), and Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS in cm). A lower score indicates less disease activity. Change from Baseline is computed as value at Week 28 minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was done using a Mixed Effects Repeated Measures Model (MMRM).
Time Frame: Baseline, Week 28
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 840
units on a scale | -21.66 (0.533)

31. Secondary Outcome: DAS28(CRP) [Disease Activity Score-28 (C-reactive Protein)] Remission (<2.6) at Week 28
Description: DAS28(CRP) is calculated using tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/L), and Patient's Global Assessment of Arthritis-Visual Analog Scale (PtGADA-VAS in mm). A lower score indicates less disease activity. This analysis was carried out using imputation.
Time Frame: Week 28
Population: Since imputation was used, all 954 subjects from the Open Label (OL) Set are included in this analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 954
percentage of subjects | 22.6

32. Secondary Outcome: SDAI (Simplified Disease Activity Index) Remission (≤3.3) at Week 28
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/dL), Patient's Global Assessment of Arthritis-Visual Analog Scale (PtGADA-VAS in cm), and Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS in cm). A lower score indicates less disease activity. This analysis was carried out using imputation.
Time Frame: Week 28
Population: Since imputation was used, all 954 subjects from the Open Label (OL) Set are included in this analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 954
percentage of subjects | 11.4

33. Secondary Outcome: CDAI (Clinical Disease Activity Index) Remission (≤2.8) at Week 28
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Arthritis-Visual Analog Scale (PtGADA-VAS in cm), and Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS in cm). A lower score indicates less disease activity. This analysis was carried out using imputation.
Time Frame: Week 28
Population: Since imputation was used, all 954 subjects from the Open Label (OL) Set are included in this analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 954
percentage of subjects | 12.1

34. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) at Week 28
Description: TJC is calculated based on tenderness response of 28 joints. TJC possible values range from 0 to 28. A lower TJC indicates less joint tenderness. Change from Baseline is computed as the value at Week 28 minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was done using a Mixed Effects Repeated Measures Model (MMRM).
Time Frame: Baseline, Week 28
Population: Of the 954 subjects in the Open Label Set (OLS) 861 had observed values at Week 28 and Baseline and are included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 861
units on a scale | -8.6 (0.26)

35. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) at Week 28
Description: SJC is calculated based on swelling response of 28 joints. SJC possible values range from 0 to 28. A lower SJC indicates less joint swelling. Change from baseline is computed as the value at Week 28 minus the baseline value. A negative value in change from baseline indicates an improvement. This analysis was done using a Mixed Effects Repeated Measures Model (MMRM).
Time Frame: Baseline, Week 28
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 861
units on a scale | -7.2 (0.19)

36. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 28
Description: HAQ-DI is derived based on the mean of individual scores in 8 categories of daily living actives (using 20 questions). Each question is scored 0-3 (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do). Change from baseline is computed as the value at Week 28 minus the baseline value. A negative value in change from baseline indicates an improvement. This analysis was done using a Mixed Effects Repeated Measures Model (MMRM).
Time Frame: Baseline, Week 28
Population: Of the 954 subjects in the Open Label Set (OLS) 854 had observed values at Week 28 and Baseline and are included in this analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 854
units on a scale | -0.46 (0.023)

37. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) at Week 28
Description: Change from Baseline in CRP (mg/L) is computed as the ratio of the value at Week 28 divided by Baseline value. A ratio less then 1 indicates an improvement. This analysis was done using a Mixed Effects Repeated Measures Model (MMRM).
Time Frame: Baseline, Week 28
Population: Of the 954 subjects in the Open Label Set (OLS) 851 had observed values at Week 28 and Baseline and are included in this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 851
mg/L | 0.59 (122.929) [0.55 to 0.63]

38. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS) at Week 28
Description: Change from Baseline in PAAP-VAS (0 to 100 mm visual analog scale, 0 being no pain and 100 being most severe pain) is computed as the value at Week 28 minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was done using a Mixed Effects Repeated Measures Model (MMRM).
Time Frame: Baseline, Week 28
Population: Of the 954 subjects in the Open Label Set (OLS) 856 had observed values at Week 28 and Baseline and are included in this analysis
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 856
mm | -23.1 (1.06)

39. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS) at Week 28
Description: Change from Baseline in PtGADA-VAS (0 to 100 mm visual analog scale, 0 being no symptoms and 100 being severe symptoms) is computed as the value at Week 28 minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was done using a Mixed Effects Repeated Measures Model (MMRM).
Time Frame: Baseline, Week 28
Population: Of the 954 subjects in the Open Label Set (OLS) 857 had observed values at Week 28 and Baseline and are included in this analysis
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 857
mm | -23.0 (1.04)

40. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS) at Week 28
Description: Change from Baseline in PhGADA-VAS (0 to 100 mm visual analog scale, 0 being no symptoms and 100 being severe symptoms) is computed as the value at Week 28 minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was done using a Mixed Effects Repeated Measures Model (MMRM).
Time Frame: Baseline, Week 28
Population: Of the 954 subjects in the Open Label Set (OLS) 848 had observed values at Week 28 and Baseline and are included in this analysis
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Open Label Certolizumab Pegol (CZP)
Number analyzed (Participants) | 848
mm | -35.6 (0.85)

ADVERSE EVENTS:
Time Frame: The first two columns refer to the 12-week double blind phase, and an additional 12-week follow up for those who withdrew during the double blind period. The third column displays AEs for the 56-week open label phase and the 12-week safety follow-up.
Description: Of the 1063 subjects in the Full Analysis Set (FAS), 1055 are included in the adverse event reporting based upon the Safety Set (SS) population. The Safety Set includes all subjects randomized who received at least 1 dosing.
Groups:
- Certolizumab Pegol (CZP): 400 mg CZP given as two 200 mg subcutaneous (sc) injections at Weeks 0, 2, and 4, followed by 200 mg CZP given as 1 sc injection on Weeks 6, 8, and 10. From Week 12, 200 mg CZP given every other week for a minimum 16 additional weeks until CZP is commercially available.
- Placebo: Placebo (0.9% saline) given as 2 subcutaneous (sc) injections at Weeks 0, 2, and 4, followed by placebo given as 1 sc injection on Weeks 6, 8, and 10. From Week 12, 200 mg certolizumab pegol (CZP) given as 1 subcutaneous injection every other week for a minimum 16 additional weeks until CZP is commercially available.
Arm/Group | Certolizumab Pegol (CZP) | Placebo | Open Label Certolizumab Pegol (CZP)
Serious Adverse Events (participants affected / at risk) | 52/846 | 12/209 | 77/954
Other Adverse Events (participants affected / at risk) | 174/846 | 42/209 | 246/954
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (CZP) (N=846) | Placebo (N=209) | Open Label Certolizumab Pegol (CZP) (N=954)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (3) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Bronchopulmonary aspergillosis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 5 (5)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 3 (4)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1) | 8 (8)
Pneumonia necrotising (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Artial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Perocardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1)
Necrosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear lobe infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Gastritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Device breakage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Polytraumatism (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian granulosa-theca cell tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Plural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Drug eurption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Synoviorthesis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Femoral arterial stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (3)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (CZP) (N=846) | Placebo (N=209) | Open Label Certolizumab Pegol (CZP) (N=954)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 37 (46) | 16 (18) | 68 (83)
Headache (Nervous system disorders) | 46 (57) | 11 (13) | 35 (40)
Upper respiratory tract infection (Infections and infestations) | 62 (68) | 11 (12) | 76 (83)
Nasopharyngitis (Infections and infestations) | 27 (31) | 4 (4) | 53 (58)
Urinary Tract Infection (Infections and infestations) | 24 (28) | 9 (10) | 64 (76)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.